CLINICAL TRIAL: NCT06233669
Title: An Analysis of Burnout Among Surgery Residents at a Tertiary Care Hospital in Pakistan
Brief Title: An Analysis of Burnout Among Surgery Residents at a Tertiary Care Hospital in Pakistan: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Mansoor Ahmed, Principal Investigator, Shaheed Zulfiqar Ali Bhutto Medical University
Other Study IDs: F.3-1/2023(ERRB)/Chairman
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Burnout, Psychological
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of Burnout — No intervention used.

SUMMARY:
To determine the scores of exhaustion, depersonalization and personal achievement according to Maslach Burnout Inventory (MBI) in surgical residents.

DETAILED DESCRIPTION:
A prospective cohort study was conducted at Pakistan Institute of Medical Sciences Islamabad with a 6-month duration from June 1, 2023 to November 30, 2023 after approval from the Institutional review board, 95 surgical residents working in Departments of Surgery & Allied of age less than 35 years (any gender) with duty of at least 60 hours per week were enrolled in study by using non-probability convenience sampling technique. Residents were informed about the study procedure and consent for inclusion was taken from them. Data analysis was done through SPSS v.26.

ELIGIBILITY:
Inclusion Criteria:

* Residents working in departments of surgery and allied
* Both genders
* Less than 35 years old
* Performing duty of at least 60 hours per week

Exclusion Criteria:

* Those who did not wish to participate

Max Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Post graduate residents working in surgery and allied.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
To determine the scores of exhaustion, depersonalization and personal achievement according to Maslach Burnout Inventory (MBI) in surgical residents. | 6 months
  These components are added to get the total score. It is interpreted as given below:
  A.Burnout i.≤ 17: Low-level burnout ii.18 to 29: Moderate burnout iii.> 30: High-level burnout B.Depersonalization i.≤ 5: Low-level burnout ii.6 to 11: Moderate burnout iii.≥ 12: High-level burnout C.Personal achievement i.≤ 33: High-level burnout ii.34-39: Moderate burnout iii.≥ 40: Low level burnout

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University/PIMS, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
Confidentiality